CLINICAL TRIAL: NCT00937989
Title: Patient Navigation in Breast Cancer Care; Addressing Barriers to Treatment Initiation, Completion, and Follow Up
Brief Title: Study of Barriers to Beginning and Finishing Treatment for Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 08092; P30CA033572 (NIH); CHNMC-08092; CDR0000629952 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; lobular breast carcinoma in situ; male breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms, Male | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: educational intervention — Occurs weekly during the first 8 weeks of the study and thereafter a minimum of monthly through the 9th month of the study.
Other: informational intervention — Occurs weekly during the first 8 weeks of the study and thereafter a minimum of monthly through the 9th month of the study.
Other: medical chart review — Baseline, 3, 6 and 9 months after starting the study
Other: questionnaire administration — Baseline, 3, 6 and 9 months after starting the study
Other: study of socioeconomic and demographic variables — Baseline, 3, 6 and 9 months after starting the study
Procedure: quality-of-life assessment — Baseline, 3, 6 and 9 months after starting the study

SUMMARY:
RATIONALE: Gathering information about barriers to receiving breast cancer treatment may help doctors learn more about improving the treatment process and improve patients' quality of life.

PURPOSE: This clinical trial is studying barriers to beginning and finishing treatment for patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify barriers of receiving primary breast cancer treatment for older patients with either Medi-Cal insurance or who are 65 years of age and older.
* Describe steps and processes involved in resolution of barriers to receiving primary breast cancer treatment for these patients.
* Identify barriers of receiving primary breast cancer treatment for patients who are Hispanic with either Medi-Cal insurance or aged 65 years and older.
* Describe steps and processes involved in resolution of barriers to receiving primary breast cancer treatment for these Hispanic patients.
* Describe breast cancer participants' perceptions of Patient Navigation.
* Demonstrate the significant role of a Patient Navigator in identifying and resolving barriers to treatment.
* Increase opportunities for participation of breast cancer patients with either Medi-Cal insurance or who are 65 years of age and older, or who are Hispanic, to breast cancer clinical trials.
* Integrate a patient navigation program within City of Hope designed to support underserved patients during primary treatment for breast cancer.

OUTLINE: For the first 3 months of the study, medical charts are reviewed.

Beginning in month 4, patients are introduced to the Patient Navigator who provides them with telephone and e-mail contact on an Appointment Reminder Card, and develops a plan for eliminating identified barriers and/or addressing immediate concerns. Patients' plans may include contacting others on behalf of the patient, coaching the patient on how to solve a problem, referring to resources within City of Hope (COH) or in the community, and investigating possible solutions. Patients are also oriented to COH's services, open clinical trials, and resources. Navigation of care includes assistance during initial and ongoing evaluations by all cancer specialists, during initiation and completion of all primary treatment, and through the first post-treatment follow up. Patients are contacted weekly for 8 weeks of the study and at least once a month for 9 months.

The Patient Navigator will track identified barriers, processes to resolution, and time required to resolve barriers.

Patients complete questionnaires at baseline, and periodically during study, on socio-demographic, quality of life, resource-use satisfaction, and satisfaction with care and Patient Navigator.

After completion of study intervention, patients continue to receive Patient Navigator support for up to 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed breast cancer

  * Stage 0-III disease
  * No metastasis or recurrent disease
* Insured with Medi-Cal OR ≥ 65 years old
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* English or Spanish-speaking
* Intending to receive all primary breast cancer treatment at City of Hope

PRIOR CONCURRENT THERAPY:

* No prior therapy for breast cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Barrier resolution (information, transportation, appointments, and communication) and time to resolution | Weekly during the first 8 weeks of the study and thereafter a minimum of monthly through the 9th month of the study.
Quality of life (psychological, physical, social, and spiritual well-being) | Prior to starting treatment and 3, 6 and 9 months after starting the study.
Navigation and care (patient's satisfaction and value, provider's perception of barriers) | 3, 6 and 9 months after starting the study.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Crane-Okada, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States